CLINICAL TRIAL: NCT03229005
Title: Influence of Soft Tissue Width and Abutment Height on Peri-implant Bone Resorption: a Clinical and Radiographic Multicenter Study
Brief Title: Soft Tissue Width and Abutment Height Influence Peri-implant Bone Resorption
Acronym: i-RES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Piezosurgery Academy (Other)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, President of the Academy, International Piezosurgery Academy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: i-RES
Record Dates: First submitted 2017-07-22; First posted 2017-07-25 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Alveolar Bone Loss
Keywords: soft tissue; implant; abutment;
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1 thick-high (Active Comparator): group with thick tissue and high prosthetic abutment tissue measurement implant insertion operculectomy prosthetic rehabilitation
  Interventions: Procedure: implant insertion; Procedure: operculectomy; Procedure: prosthetic rehabilitation
- A2 thick-low (Experimental): group with thick tissue and low prosthetic abutment tissue measurement implant insertion operculectomy prosthetic rehabilitation
  Interventions: Procedure: implant insertion; Procedure: operculectomy; Procedure: prosthetic rehabilitation
- B1 thin-high (Active Comparator): group with thin tissue and high prosthetic abutment tissue measurement implant insertion operculectomy prosthetic rehabilitation
  Interventions: Procedure: implant insertion; Procedure: operculectomy; Procedure: prosthetic rehabilitation
- B2 thin-low (Experimental): group with thin tissue and low prosthetic abutment tissue measurement implant insertion operculectomy prosthetic rehabilitation
  Interventions: Procedure: implant insertion; Procedure: operculectomy; Procedure: prosthetic rehabilitation

INTERVENTIONS:
Procedure: implant insertion — during surgery soft tissues will be measured
Procedure: operculectomy — during second surgery soft tissues will be measured again
Procedure: prosthetic rehabilitation — after three months implants will be loaded with screw retained crown

SUMMARY:
The purpose of this clinical and radiographic study will be to determine what influence on marginal bone loss has the thickness of soft tissues and the height of the prosthetic abutment and eventually determine which of the two factors is the most important.This research was designed as a multicentre cohort study. Two clinical centers will treat patients through the placement of a single dental implant. The implants will be prosthetically loaded about 4 months after placement and periapical radiographs will be acquired at each time-point.

DETAILED DESCRIPTION:
The purpose of this clinical and radiographic study will be to determine what influence on marginal bone loss has the thickness of soft tissues and the height of the prosthetic abutment and eventually determine which of the two factors is the most important.This research was designed as a multicentre cohort observational study. Two clinical centers will treat patients through the placement of a single dental implant. The implants will be prosthetically loaded about 4 months after placement and periapical radiographs will be acquired at each time-point.

All patients will receive antibiotic prophylaxis with 2 g of amoxicillin one hour before surgery. With the help of a dissector, a full thickness vestibular flap will be carefully arranged and the vertical thickness of soft tissues will be measured with a probe marked every 1.0 mm. If the vertical thickness of the soft tissue is 2 mm or less, the tissue will be considered thin. If the thickness of the mucosa is greater than 2 mm, it will be considered thick. After the measurement, the lingual flap will be elevated at full thickness, and the site for site placement will be prepared. The implant bed will be at least 1.5 mm from the adjacent tooth or teeth, and must be surrounded by at least 1 mm bone in both buccal and lingual directions. A 3,75 mm diameter and internal hexagonal connection implant will be placed at the level of the bone crest according to the manufacturer's recommendations. Operators will be free to choose the most suitable system length (8, 10, 11.5 mm). All implants will be submerged according to a traditional two-stage protocol. After insertion, the flaps will be sutured without tension with interrupted sutures. Patients of both groups will be instructed to disinfect the site by rinsing twice daily for one week for 1 minute with 0.12% chlorhexidine. After 4 months of healing, the treated area will be reopened for connecting the healing abutments with a crestal incision that will retain the keratinized tissue; The same soft tissue measurements will be repeated as confirmation of what was done during the first surgical implant insertion phase. The implants will be considered osteointegrated successfully if they are clinically intact unless they show obvious radiotransparency and patients will not report any pain. After this step, it will be possible to divide the patients into 2 groups according to the thickness of the soft tissue: a group with thick tissue (more than 2.0 mm); Slim tissue group (less than 2.0 mm). The prosthetic framework will be bonded directly to prefabricated titanium abutment (1 or 3 mm). This will result in the formation of 4 different subgroups: a group with thick tissue and high prosthetic abutment; A group with thick tissue and low prosthetic stump; a group with thin tissue and high prosthetic abutment; a group with thin tissue and low prosthetic abutment.

All the implants will be rehabilitated by the dentist with screwed restorations. After prosthetic treatment, patients will receive oral hygiene instructions and will be monitored through calls to ensure periodontal health throughout the study period.

ELIGIBILITY:
General inclusion criteria were:

* age>18 years;
* good general health;
* non smokers;
* absence of systemic diseases affecting bone metabolism and wound healing; - no regular medication consumption for at least 3 months prior to treatment; - patient willing and fully capable to comply with the study protocol;
* written informed consent given.

Local inclusion criteria were:

* presence of keratinized mucosa with a minimum bucco-lingual width of 3 mm; - bone crest with at least 6 mm of width and 9 mm of height above the mandibular canal, without concomitant or previous bone augmentation procedures;
* presence of the opposing dentition.

Exclusion criteria were:

* history of head or neck radiation therapy;
* uncontrolled diabetes (HBA1c >7.5%);
* active infections;
* immunocompromised patients (HIV infection or chemotherapy within the past 5 years);
* present or past treatment with intravenous bisphosphonates;
* patient pregnancy or lactating at any time during the study;
* poor oral hygiene and motivation;
* untreated periodontal disease;
* psychological or psychiatric problems;
* alcohol or drugs abuse;
* participating in other studies, if the present protocol could not be properly followed;
* lack of implant primary stability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
peri-implant bone resorption | after 12 months
  intraoral radiographs will be acquired and bone crest level will be compared with baseline
implant survival | after 12 months
  clinical and radiographical examination

SECONDARY OUTCOMES:
peri-implant bone resorption | immediately after surgery (baseline)
  intraoral radiographs will be acquired
peri-implant bone resorption | four months after surgery (at prosthesis delivery)
  intraoral radiographs will be acquired
peri-implant bone resorption | six months after prosthetic loading
  intraoral radiographs will be acquired
peri-implant bone resorption | 24 months after prosthetic loading
  intraoral radiographs will be acquired
complications and/or adverse events | any time of the study
  clinical and radiographical examination

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr., Principal Investigator — Piezosurgery Academy
Locations (1):
- Piezosurgery Academy, Parma, PR, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galindo-Moreno P, Leon-Cano A, Monje A, Ortega-Oller I, O'Valle F, Catena A. Abutment height influences the effect of platform switching on peri-implant marginal bone loss. Clin Oral Implants Res. 2016 Feb;27(2):167-73. doi: 10.1111/clr.12554. Epub 2015 Feb 11. PMID 25678247
- [Background] Linkevicius T, Apse P, Grybauskas S, Puisys A. Influence of thin mucosal tissues on crestal bone stability around implants with platform switching: a 1-year pilot study. J Oral Maxillofac Surg. 2010 Sep;68(9):2272-7. doi: 10.1016/j.joms.2009.08.018. PMID 20605308